CLINICAL TRIAL: NCT03424837
Title: Evaluation of the Impact of A Survivorship Care Plan and Embedded Navigation Tool (ASCENT) in Patients With Prostate Cancer Undergoing Curative-Intent Radiotherapy With Concurrent Androgen Deprivation Therapy (ADT)
Brief Title: A Survivorship Care Plan and Embedded Navigation Tool
Acronym: ASCENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of Michigan (Other); Emory Healthcare (Other); Johns Hopkins University (Other); Memorial Sloan Kettering Cancer Center (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); UNC Lineberger Comprehensive Cancer Center (Other); Morehouse School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00088754
Record Dates: First submitted 2018-01-26; First posted 2018-02-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: SoC (standard of care) and ASCENT (Experimental): Health care per institutional standard plus ASCENT via the TrueNTH website.
  Interventions: Behavioral: ASCENT
- Control Arm: SoC and TrueNRH (No Intervention): Health care per institutional standard, plus access to the public information on the TrueNTH website; such as the symptom tracker, exercise & diet, and lived experiences modules.

INTERVENTIONS:
Behavioral: ASCENT — ASCENT includes the following components:
  * Survivorship care plan created through the ASCENT tool
  * Online tool which assesses health care needs and facilitates receipt of care
  * A national-level navigator who helps the participant to access support services
  * Periodic reminders for the participant to pursue recommended survivorship care
  Arms: Intervention Arm: SoC (standard of care) and ASCENT

SUMMARY:
This is a parallel group, multisite prospective clinical study. The purpose of this study is to evaluate whether ASCENT enables patients to adhere to the survivorship guidelines and improves coordination of care to address patient needs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of prostate adenocarcinoma
* Age ≥18 years
* Receiving curative intent radiotherapy for prostate cancer (Note: post-operative radiotherapy [i.e., "adjuvant" or "salvage radiotherapy subsequent to prostatectomy] is allowed.)
* Subjects will be enrolled within two weeks prior to and two weeks after the final fraction of radiotherapy.
* Receiving androgen deprivation therapy (ADT) for a duration of ≥3 consecutive months as follows:

  * GnRH agonist or antagonist (medical castration), with or without an anti-androgen (i.e., bicalutamide, flutamide, nilutamide, etc.), OR
  * Bilateral orchiectomy (surgical castration)
* Technology requirement: candidates must have access to the internet
* Able to understand and willing to sign a written informed consent document.
* Able to speak and understand English, in the opinion of the treating physician.

Exclusion Criteria:

* Significant concurrent medical or psychiatric condition that would interfere with the patient's ability to abide by the study protocol or cooperate fully with the protocol requirements, including completion of survey and assessment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2020-11-24 (Actual); Study Completion 2020-11-24 (Actual)

PRIMARY OUTCOMES:
Abiding by the survivorship guidelines as measured by making an appointment within 6 months of enrollment OR completing a guideline-based assessment. | 6 months
  Abiding by the survivorship guidelines is defined as either of: Making an appointment with primary health care provider within 6 months of enrollment, OR completing a guideline-based assessment or management strategy for reducing side effects related to prostate cancer treatment.
Assess trial participants', caregivers'/family members', and staff satisfaction and experiences with the ASCENT technology and trial. | 6 months
  Focus group comments and question responses detailing trial participants', caregivers'/family members', and staff's satisfaction and experiences with ASCENT.

SECONDARY OUTCOMES:
General health status | 6 months
  General health status will be measured using the EuroQol five dimensions questionnaire (EQ-5D).
Existence and severity of depression | 6 months
  Existence and severity of depression will be evaluated using the Patient Health Questionnaire (PHQ-9).
Prostate-cancer specific quality of life. | 6 months
  Prostate-cancer specific quality of life will be determined using the Expanded Prostate Cancer Index Composite - Short Form (EPIC-26).
Overall health-related-quality of life including, but not limited to, mental and physical functioning as measured by the Short Form Health Survey | 6 months
  Overall health-related-quality of life will be measured using the Short Form Health Survey (SF-12).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harrison, M.D., Principal Investigator — Duke University; Andrew Peterson, M.D., Principal Investigator — Duke University
Locations (6):
- United States (6):
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University & Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins School of medicine & Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Cancer Center, Chapel Hill, North Carolina
  - Duke Cancer Institute, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No